CLINICAL TRIAL: NCT06800482
Title: A Randomized Controlled Study of Online Outpatient Follow-up in Patients With Papillary Thyroid Cancer After Surgery
Brief Title: A Study of Online Follow-up in Patients With Papillary Thyroid Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xinyi Wang, Principal Investigator, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: WestChinaH20241018
Record Dates: First submitted 2024-11-28; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Thyroid; Papillary Thyroid Cancer
Keywords: Papillary thyroid cancer; surgery; out-patient
MeSH Terms: conditions — Thyroid Diseases; Thyroid Cancer, Papillary

STUDY DESIGN:
Intervention Model Description: Using the REDCap randomization module, a computer-generated permutation block randomization, with random block sizes of 6 and 9, randomly assigned participants to online or offline visits in a 1:1 manner. The assignment order is hidden, and the results of the post-assignment randomization are extracted by an independent data collection team. Participants who visit online are given a booklet detailing how to access the platform and create a secure login and a phone number to schedule an appointment. Participants who do not call within 3 working days of the expected follow-up time after discharge will be called up to 2 times by the outpatient assistant to schedule an appointment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Using Huayitong APP in participants with papillary thyroid cancer (Active Comparator): Post-operative follow-up was performed using Huayitong APP
  Interventions: Behavioral: online outpatient follow-up
- standard offline outpatient follow-up in patients with papillary thyroid cancer (No Intervention): Participants were followed up in traditional offline outpatient clinics

INTERVENTIONS:
Behavioral: online outpatient follow-up — The investigators use Huayitong APP for the post-operating follow-up of participants with papillary thyroid cancer
  Arms: Using Huayitong APP in participants with papillary thyroid cancer

SUMMARY:
The randomized, actively controlled, non-inferiority trial is scheduled to begin in August 2024 and run through August 2026. Inclusion criteria: (1) has undergone microwave ablation of thyroid or thyroidectomy (including endoscopy and opening) at the Department of Thyroid Surgery of West China Hospital of Sichuan University, (2) is between 18 and 90 years old, (3) speaks Chinese, (4) has the email address and operational ability required to complete the visit, (5) does not have a mental illness or take psychotropic drugs, (6) Voluntarily participate in clinical trials and sign informed consent. Exclusion criteria: (1) postoperative hospital stay more than 3 days; (2) Inability to complete an online visit (no access to the device or the Internet); (3) High risk of postoperative complications (recurrent laryngeal nerve injury, etc.); (4) Inability to participate due to a medical condition, laboratory test results, or physical disability (as determined by the principal investigator or surgeon).

The online outpatient follow-up was completed by thyroid surgeons of West China Hospital. Informed consent signed with a voluntary participant after a research team member contacts the patient and introduces the patient to the study. The investigators who contacted, enrolled, and randomly assigned patients included the principal investigator, the study coordinator, and the research assistant who had been specially trained in the study.

According to the agreement, the participants randomly assigned to online visits will cross over with offline visits and withdraw from the clinical trial if :(1) unresolved technical issues, (2) inability to perform a full evaluation, (3) need/request prescription painkillers, and (4) additional care recommended by a physician. Other cross-cutting reasons include patient requests and scheduling conflicts.

The information department of WestChina hospital obtained online and offline participants' demographic data and comorbidities, related information of chief complaint (including time of illness, information of last visit, drugs being used, contents of consultation, disease symptoms, conclusions of consultation, etc.), and online and offline outpatient information (including application time, reception time, patient satisfaction, etc.). Whether to prescribe medicine, whether to prescribe examination/admission certificate, outpatient cost, number of questions, number of return visits, etc.) Employment, living conditions and the highest education level were obtained through the questionnaire survey at the time of enrollment, and the information about participant experience and satisfaction was obtained through the questionnaire survey after follow-up. The investigators recorded the diagnosis and treatment details of the patients at three online/offline follow-up visits at 1, 3, and 6 months after surgery. The investigators reviewed the electronic medical record 30 days after the last follow-up to monitor for adverse events. Participants were surveyed by email 30 days after the last follow-up to assess adverse events, including readmissions. If the survey is not answered within a week, an electronic reminder is sent and two attempts are made to contact the participants by phone.

ELIGIBILITY:
Inclusion Criteria：

* clinical diagnosis of papillary thyroid cancer
* has underwent thyroid surgery (including endoscopic and open thyroid surgery)
* 18 to 90 years of age
* spoke Chinese
* has the ability to use mobile phones and the Internet to complete the visit
* voluntarily participate in clinical trials and sign informed consent.

Exclusion Criteria：

* postoperative hospital stay more than 5 days
* inability to complete an online visit (no access to the device or the Internet
* high risk of postoperative complications (recurrent laryngeal nerve injury, etc.)
* unable to participate due to comorbidities, laboratory test results or physical disability
* pregnancy
* has mental illness or take psychotropic drugs, and were not able to perform the surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 388 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
The adherence to outpatient procedures | From enrollment to the end of follow-up at 12 months
  At 12 months after the operation, the participants' medical information is extracted through the electronic recording system of Huatong APP to determine whether the participants complied with the random group for postoperative follow-up. The data were extracted by the Information Department of West China Hospital.

SECONDARY OUTCOMES:
General life quality of participants | From enrollment to the end of follow-up at 12 months
  Questionnaire assessment for each assessment time point will be conducted in the thyroid surgery ward of West China Hospital of Sichuan University. Before each assessment time point, the investigators will notify the participants in advance by phone or wechat and inform them of relevant precautions. Participant's life qualities are measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTCQLQ-C30), referring to the following articles: PMID: 36376888, PMID: 34985562.

OTHER OUTCOMES:
Thyroid related symptom score | From enrollment to the end of follow-up at 12 months
  Questionnaire assessment for each assessment time point will be conducted by study participants in the thyroid surgery ward of West China Hospital of Sichuan University. Before each assessment time point, the investigators will notify the participants in advance by phone or wechat and inform them of relevant precautions.
  Thyroid related symptom scores are measured by the thyroid cancer-specific quality of life questionnaire (THYCA-QoL), referring to the following articles: PMID: 33896584, PMID: 23013266.
Participants's satisfacation | From enrollment to the end of follow-up at 12 months
  Questionnaire assessment for each assessment time point will be conducted by study participants in the thyroid surgery ward of West China Hospital of Sichuan University. Before each assessment time point, the investigators will notify the participants in advance by phone or wechat and inform them of relevant precautions. Participant's satisfaction with the doctor are granded from 1 to 10, with 1 is the least satisfied and 10 is the most satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China